CLINICAL TRIAL: NCT07207083
Title: Effects of Immersive Virtual Reality-based Exercise on Somatosensory Function, Pain, and Psychological and Functional Recovery in Patients With Chronic Low Back Pain
Brief Title: Can Virtual Reality Exercise Help Restore Both Body and Mind in Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: dongmin kang (Other)
Responsible Party: Sponsor-Investigator, dongmin kang, Master's Degree Candidate, Sahmyook University
Organization: Sahmyook University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYU 2025-08-019-002
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Virtual Reality; Kinesiophobia; Chronic Low Back Pain (CLBP); Central Sensitization; Fear of Movement
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. The experimental group will perform immersive Virtual Reality-based exercise using the FitXR application, while the control group will perform the same exercise protocol without VR immersion. Both groups will receive 15-minute exercise sessions over the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Exercise Group (Experimental): Participants perform a 15-minute exercise program using immersive virtual reality (FitXR app with Meta Quest 3s).
  Interventions: Behavioral: Immersive Virtual Reality-based Exercise (FitXR, Meta Quest 3s)
- Non-VR Exercise Group (Active Comparator): Participants perform the same 15-minute exercise program, but without VR equipment.
  Interventions: Behavioral: Conventional Exercise Program (Matched Exercise, without VR)

INTERVENTIONS:
Behavioral: Immersive Virtual Reality-based Exercise (FitXR, Meta Quest 3s) — participants assigned to the intervention group will perform a 15-minute immersive virtual reality (VR) exercise program using the FitXR application on the Meta Quest 3s headset.
  This program provides interactive, visually immersive exercise tasks designed to engage participants in physical activity while reducing fear of movement and enhancing functional recovery.
  Arms: VR Exercise Group
Behavioral: Conventional Exercise Program (Matched Exercise, without VR) — Participants assigned to this arm will perform the same 15-minute exercise program without virtual reality equipment.
  This allows comparison between immersive VR-based exercise and conventional exercise of equivalent intensity and duration.
  Arms: Non-VR Exercise Group

SUMMARY:
The goal of this clinical trial is to learn if an immersive virtual reality (VR) exercise program can help reduce back pain and improve physical function and psychological well-being in adults with chronic low back pain.

The main questions it aim to answer are

* Does the virtual reality (VR) exercise reduce back pain?
* Does it lead to positive changes in how participants perceive pain?
* Does it improve back flexibility and reduce disability in daily activities?
* Does it help reduce the fear of movement and negative thoughts related to pain? Method Wear a Meta Quest 3s device and participate in a 15-minute virtual reality exercise program called 'FitXR'.

Be evaluated for their back pain, sensory test, range of motion, and level of disability in daily life before and after the exercise program.

Complete questionnaires about their thoughts and feelings regarding their pain and movement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* Non-specific chronic low back pain lasting ≥3 months.
* Baseline pain intensity VAS ≥4/10.
* Kinesiophobia (TSK-13) ≥34.
* Able to perform physical activity using immersive VR (screened as suitable for head-mounted display-based activity).
* Understands the study purpose and procedures and provides written informed consent.

Exclusion Criteria:

* Severe pain making participation infeasible: VAS ≥8/10.
* Lumbar spine surgery within the past 6 months.
* Severe musculoskeletal disorders (e.g., advanced osteoarthritis, pathological vertebral fracture).
* Neurological disorders (e.g., multiple sclerosis, Parkinson's disease, stroke).
* Cardiovascular disease (e.g., heart failure, clinically significant arrhythmia, recent myocardial infarction).
* Simulator Sickness Questionnaire (SSQ): total score ≥20 or any single item scored 3.
* Vulnerable populations excluded: minors, older adults, individuals with psychiatric disorders or cognitive impairment, and pregnant persons.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST): Specifically including Conditioned Pain Modulation (CPM) and Temporal Summation (TS) protocols. | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  CPM measures the efficiency of the body's pain-inhibiting pathways. A higher positive value indicates a more effective pain modulation system (better outcome). TS measures pain sensitization. A higher score indicates greater central sensitization to pain (worse outcome).

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia-13 (TSK-13) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  The scale scores range from 13 to 52. A higher score indicates a greater degree of kinesiophobia (fear of movement), which is a worse outcome.
Pain Catastrophizing Scale (PCS) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  The scale score ranges from 0 to 52. A higher score indicates a greater level of pain catastrophizing (a worse outcome).
Oswestry Disability Index (ODI) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  This index measures disability due to low back pain, with the score reported as a percentage from 0% to 100%. A score of 0% indicates no disability, while 100% indicates the most severe disability (a worse outcome).
Fear-Avoidance Beliefs Questionnaire (FABQ) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  This questionnaire has two subscales: Physical Activity (range 0-24) and Work (range 0-42). For both scales, a higher score indicates stronger fear-avoidance beliefs (a worse outcome).
Visual Analog Scale (VAS) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  This scale measures the intensity of pain. It is typically a 100-millimeter line on which participants mark their pain level. A score of 0 mm indicates "no pain", while 100 mm indicates "the worst pain imaginable". A lower score represents a better outcome.
Lumbar Range of Motion (ROM) | Measured at Week 1 (baseline), Week 6 (post-intervention), and Week 8 (follow-up).
  This is a physical measurement of lumbar spine flexibility, objectively assessed using a dual inclinometer. The range of motion for flexion, lateral bending is reported in degrees (°). A higher value, representing a greater range of movement, indicates better physical function (a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Science Hall 3, Seoul, Seoul, South Korea